CLINICAL TRIAL: NCT00491660
Title: Effect of Gravity on Tracheal Colonization During Mechanical Ventilation in Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2004-MD-Thesis-Afaf
Record Dates: First submitted 2007-06-25; First posted 2007-06-26 (Estimated); Last update posted 2007-06-26 (Estimated); Status verified 2007-06

CONDITIONS: Pneumonia, Ventilator-Associated
Keywords: Gravity; Mechanical ventilation; Infants; Ventilator-associated pneumonia; Types of bacterial colonies in subjects at 2-5 days of mechanical ventilation; Colony count of an organism was cultured
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

INTERVENTIONS:
Behavioral: supine positioning
Behavioral: lateral positioning

SUMMARY:
Ventilator-associated pneumonia (VAP) is the leading cause of death among all nosocomial infections in ventilated patients. Once intubated, the risk of pneumonia in hospitalized patients is increased 3-10 fold; almost 90% of hospital-acquired pneumonia occurs in intubated patients. Each episode of VAP is associated with 7-9 days of additional hospital stay with an estimated increase in cost of care that exceeds $40,000. In an effort to control VAP, several studies were conducted including oral and gastric decontamination with antibiotics, rotation of the bed, and local instillation of antibiotics via endotracheal tube. Despite such efforts, VAP is still a major complication for intubated patients.

The effect of gravity on bacterial colonization of the endotracheal tube was recently explored in an animal study that was conducted at the United States National Institutes of Health. The study demonstrated a significantly lower tracheal colonization and decreased alveolar contamination in ventilated sheep when positioned on their side allowing for tracheal drainage by gravity. Such findings have not been validated in clinical practice and the need for clinical trials studying the effect of lateral positioning have been demanded. Therefore, we aimed our randomized controlled trial to test the hypothesis that intubated infants who are positioned on their side are at lower risk for contracting microbes in their trachea when compared to those in a supine position.

DETAILED DESCRIPTION:
Subjects were to be randomly assigned to one of two groups:

1. Supine group, in which infants are maintained on their back at all times. The endotracheal tube is held upright in vertical position at all times. The bed is kept horizontal without any angle or tilt.
2. Lateral group. Infants are maintained on their side while the back supported with a rolled towel. The endotracheal tube is maintained to rest horizontally on the bed.

ELIGIBILITY:
Inclusion Criteria:

* Term and premature infants >28 weeks of gestation
* Postnatal age <48 hours
* Mechanical ventilation >5 days

Exclusion Criteria:

* Congenital infections
* Congenital pneumonia
* Congenital anomalies such as tracheal-esophageal fistula, thoracic cage deformities and diaphragmatic hernia
* not maintained on mechanical ventilation for 5 complete days

Max Age: 48 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2005-01; Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Rate of colonization in tracheal aspirates at 2 days | 2 days

SECONDARY OUTCOMES:
Number of colonies in colonized infants | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Magda Badawy, MD, Study Chair — Cairo University Children's Hospital; Afaf Mohamed, M.B,B.Ch, Principal Investigator — Cairo University Children's Hospital